CLINICAL TRIAL: NCT03551379
Title: Single Center Prospective Evaluation Utilizing a Double Balloon Accessory Device to Facilitate Complex Endoscopic Polypectomy in Large Intestine
Brief Title: A Double Balloon Endoscopic Platform for ESD
Status: Completed | Type: Observational
Sponsor: Lumendi, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: DD-017
Record Dates: First submitted 2018-05-08; First posted 2018-06-11 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Colon Adenoma; Colon Polyp
Keywords: Endoscopic Submucosal Dissection
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Endoscopic procedure: A double balloon endoscopic platform will be used during an ESD procedure
  Interventions: Device: Double Balloon Endoluminal Platform

INTERVENTIONS:
Device: Double Balloon Endoluminal Platform — A DBA platform will be use din this registry study to facilitate ESD

SUMMARY:
The purpose of this observational study is to record performance of a double balloon endolumenal interventional platform during complex colon polypectomy.

DETAILED DESCRIPTION:
Endoscopic removal of Complex colon polyps (benign polyps >=2cm) is a technically challenging procedure. Complex benign polyps have a greater chance of becoming cancerous if not removed.

The DiLumen™ Endolumenal Interventional Platform is a non-sterile, single-use, close-fitting sleeve that fits securely over a standard endoscope to stabilize it in the large intestine, and facilitates use of the endoscope for optical visualization, diagnosis, and treatment. The device is indicated to ensure complete positioning of an endoscope in the large intestine and assist with optical visualization, diagnosis, and endoscopic treatment.

The device received 510k clearance on Dec 6, 2016. The study will evaluate performance of the device during routine, scheduled, endoscopic polyp removal for these large polyps.

ELIGIBILITY:
Inclusion Criteria:

* Subjects > 18 years of age
* Subjects scheduled for endoscopic removal of suspected complex adenomatous polyps in the large intestine which are sessile or polypoid lesions ≥ 2cm, near the ileocecal valve, dentate line, over a fold, or at a flexure; and or lesions tethered to the colon wall due to previous incomplete resection
* Subjects willing and able to give informed consent
* Subjects who in the opinion of the Principal Investigator have no medical contraindication to endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD)

Exclusion Criteria:

* Subjects with a contraindication to colonoscopy, including but not limited to active colitis, perforation, or stricture.
* Subjects with a history of open or laparoscopic colorectal surgery
* Subjects with a history of Inflammatory Bowel Disease (IBD)
* Subjects with a suspected malignancy on polyp assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with documented complex large intestinal polyps
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-09-29 (Actual)

PRIMARY OUTCOMES:
Ability to remove the complex polyp endoscopically | Duration of Procedure
  Was the lesion(s) able to be removed using the DiLumen Endolumenal Interventional Platform Device [Yes/No]
Time taken for lesion removal | Intervention start time until Lesion removal
  Time for lesion(s) removal with the double balloon device after intervention begins
Device or Procedural Adverse Events | Up to 72 hours
  Colon perforation, colon mucosal injury, excess bleeding will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Stavropoulos, MD, Principal Investigator — Winthrop-NYU Langone Mineola, NY
Locations (1):
- Winthrop-NYU Langone, Mineola, New York, United States

IPD SHARING:
Plan to Share IPD: No